CLINICAL TRIAL: NCT05596877
Title: The Effect of Music Therapy on Anxiety and Perceived Time in Pulmonary Rehabilitation
Brief Title: Music Therapy in Pulmonary Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Group leader of Respiratory Therapists, Fu Jen Catholic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FJUH111237
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2022-12

CONDITIONS: Chronic Pulmonary Disease
Keywords: Music therapy; Pulmonary rehabilitation; Depression; Percieved time; Chronic obstructive pulmonary disease
MeSH Terms: conditions — Depression; Pulmonary Disease, Chronic Obstructive | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Recieved pulmonary rehabilitation
- Intervention Group (Experimental): Recieved pulmonary rehabilitation with music therapy
  Interventions: Behavioral: Music therapy

INTERVENTIONS:
Behavioral: Music therapy — Performing music therapy during a course of pulmonary rehabilitation (25 mins)
  Arms: Intervention Group

SUMMARY:
This study explores the effects of music therapy intervention on anxiety and time perception during pulmonary rehabilitation.

DETAILED DESCRIPTION:
Background：

In recent years, in many domestic and foreign music therapy literature, it can be found that the intervention of music therapy can alleviate the anxiety of patients in the treatment, surgery, and even patients with critical care using ventilators, and then affect the patient's physiological indicators, in addition, there are also studies that mention that background music affects people's waiting time perception, reduces people's waiting time, can reduce the generation of negative emotions, and improve the quality of hospital medical care. The objective of this study was to explore the effects of music therapy on anxiety and time perception during pulmonary rehabilitation.

Study Design：

This case is a one-year single-center, prospective block randomizied trial.

Methods：

The study is expected to be 50 people, randomly assigned to two groups (control group, experimental group) will be carried out in the pulmonary rehabilitation room on the sixth floor of the Fu Jen Catholic University Hospital, using the Baker Anxiety Scale, physiological monitoring instruments and cardiac output monitor as tools to test the effects of anxiety sensations, physiological responses (heartbeat, breathing times, blood pressure, heart rate variability) and perceptual time in two situations of interventional music therapy and non-interventional music therapy during the rehabilitation of negative pressure respirators.

Effect：

It was mainly found that the intervention of music therapy can reduce anxiety, number of heartbeats, number of breaths and blood pressure, and shorten the perceptual time of patients with pulmonary rehabilitation.

Key words：

Music therapy; pulmonary rehabilitation; depression; percieved time; chronic obstructive pulmonary disease

ELIGIBILITY:
Inclusion Criteria:

* Recieved pulmonary rehabilitation at least three months
* Recieved a negative ventilation during a pulmonary rehabilitation
* A written informed consent

Exclusion Criteria:

* impaired of hearing
* decline to participate
* cognitive communication deficits
* acute exacerbation of copd within three months

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-02-11 (Actual); Study Completion 2023-02-11 (Actual)

PRIMARY OUTCOMES:
Beck Anxiety Inventory's score | 25 minutes
  Beck Anxiety Inventory's score (0 present as minimal and 63 present as maximal, higher scores mean a worse outcome)

SECONDARY OUTCOMES:
Respiratory rate | 25 minutes
  Respiratory rate during a course of pulmonary rehabilitation
Heart rate variability | 25 minutes
  Heart rate variability during a course of pulmonary rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, PhD, Principal Investigator — Fu Jen Catholic University Hospital
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No